CLINICAL TRIAL: NCT04184492
Title: A Randomized Double Blinded Two-way Crossover Single-dose Pharmacokinetics and Pharmacodynamics Study of GP-40081 (LLC "GEROPHARM", Russia) Versus NovoMix® 30 Penfill® (Novo Nordisk) in Healthy Subjects Using the Euglycemic Clamp Technique
Brief Title: A Study to Compare Pharmacokinetics and Pharmacodynamics of GP-40081 to NovoMix® 30 Penfill® in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GP-40081-P4-11
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Clamp Study
Keywords: Pharmacokinetics; Pharmacodynamics; Biphasic Insulin Aspart
MeSH Terms: interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Intervention Model Description: two-way crossover
Who Masked: Outcomes Assessor
Masking Description: This study was blinded for Sponsor, investigators and analytical laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP-40081 (Experimental): Single subcutaneous administration of GP-40081 in dose 0.4 IU / kg
  Interventions: Drug: GP-40081
- NovoMix® 30 Penfill® (Active Comparator): Single subcutaneous administration of NovoMix® 30 Penfill® in dose 0.4 IU / kg
  Interventions: Drug: NovoMix® 30 Penfill®

INTERVENTIONS:
Drug: GP-40081 — biphasic insulin aspart 30 in doses 0.4 IU/kg
  Other Names: biphasic insulin aspart 30
  Arms: GP-40081
Drug: NovoMix® 30 Penfill® — biphasic insulin aspart 30 in doses 0.4 IU/kg
  Other Names: biphasic insulin aspart 30
  Arms: NovoMix® 30 Penfill®

SUMMARY:
Pharmacokinetics and pharmacodynamics study of 2 formulations of biphasic insulin aspart 30 (GP-40081 GEROPHARM vers. NovoMix® 30 Penfill® Novo Nordisk)

DETAILED DESCRIPTION:
A randomized double blinded two-way crossover single-dose pharmacokinetics and pharmacodynamics study of GP-40081 (LLC "GEROPHARM", Russia) versus NovoMix® 30 Penfill® (Novo Nordisk) in normal healthy subjects using the euglycemic clamp technique

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Caucasian males having a confirmed healthy diagnosis as per data of standard clinical, laboratory, and instrumental examination methods.
3. Age of 18-45 (both incl.).
4. Body mass index equal to 18.5-30.0 kg/m2, body weight equal to 60.0-100.0 kg (both incl.).
5. Volunteers' consent to all restrictions imposed during the study, including adequate methods of contraception.
6. Russian citizenship.

Exclusion Criteria:

1. Weighed allergic anamnesis.
2. Increased sensitivity in the history of heparin, insulin or any of the excipients of the study drugs.
3. Any acute and chronic diseases (for 4 weeks before screening) incl.:

   1. of the cardiovascular system, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.
   2. positive tests: hepatitis B (Ag), hepatitis C (Ab), HIV (Ab), syphilis (Ab).
4. Deviations in basic vital signs: heart rate (60-89), systolic blood pressure (90-139 mm Hg), the diastolic blood pressure (60-89 mm Hg), respiratory rate (12-20), body temperature (35.7-37.2 C).
5. Abnormalities of the ECG from the norms.
6. Episodes of hypoglycemia in the anamnesis; the presence in the family history of cases of a verified diagnosis of diabetes mellitus in the immediate family.
7. Fasting plasma glucose> 6.1 mmol / L.
8. HbA1C> 6% (screening).
9. Oral glucose tolerance test - blood glucose level ≥ 7.8 mmol / l (2 hours after loading with glucose).
10. Deep vein thrombosis of lower extremities in a history of life or in a family history.
11. Any diet (vegetarian, etc.), extreme physical exercise, night shift work.
12. Subjects who have taken any drugs known effects on hemodynamics or to induce or inhibit hepatic drug metabolism within 2 months prior to screening.
13. Taking medications, phytopreparations, biologically active supplements less than 14 days before screening.
14. History of significant drugs abuse conditions for 3 years prior to screening.
15. Significant blood loss (450 mL or more) less than 3 months before the screening.
16. Recovery after surgery process; scheduled surgery.
17. Mental, physical and other reasons that do not allow to adequately assess their behavior and properly fulfill the conditions of the research protocol, including psychiatric disorders.
18. A positive test for the content of drugs in the urine (screening).
19. Positive test for alcohol content in the exhaled air.
20. Receiving more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of wine or 50 ml of strong alcohol) or anamnestic information about alcoholism.
21. Nicotine dependence (use of tobacco less than 6 months before the start of screening).
22. Participation in a clinical trial of any medications less than 3 months or 5 half-lives before the IP administration.
23. Any conditions that make it difficult, according to the informed opinion of the investigating physician, that volunteer participation in studies.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | -60, -30, 0 minutes (pre-dose) and 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 180, 210, 240, 270, 300, 360, 420, 480, 600, 720, 960, 1200 and 1440 minutes post-dose
  Pharmacokinetics of insulin aspart by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))
Cmax | -60, -30, 0 minutes (pre-dose) and 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 180, 210, 240, 270, 300, 360, 420, 480, 600, 720, 960, 1200 and 1440 minutes post-dose
  Pharmacokinetics of insulin aspart by Assessment of Observed Maximum Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Endocrinology Research Centre, Moscow
  - Almazov National Medical Research Centre, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No